CLINICAL TRIAL: NCT04205214
Title: A Randomised Control Trial of Integrative Cognitive Behavioural Therapy for Alopecia: A Pilot Study
Brief Title: A Randomised Control Trial of Integrative Cognitive Behavioural Therapy for Alopecia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSYETH (P/F) 17/18 177
Record Dates: First submitted 2019-11-10; First posted 2019-12-19 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-01

CONDITIONS: Alopecia
Keywords: Cognitive Behavioural Therapy; Mindfulness; Narrative Therapy; Alopecia Areata; Alopecia Universalis; Alopecia Totalis; Psychology; Health Psychology
MeSH Terms: conditions — Alopecia; Alopecia Areata; Alopecia universalis

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants are not aware of their allocation to the intervention group or control group. All
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative Cognitive Behavioural Therapy Intervention Group (Experimental): The group receive 12 weekly individual Integrative Cognitive Behavioural Therapy sessions from the principal investigator and Trainee counselling Psychologist. The sessions last up to 60 minutes on a weekly basis. The participants in this group are required to complete self-reported questionnaires assessing: anxiety, depression, stress and quality of life. They are also required to attend a scalp assessment and undergo a blood test and medical photography. These assessments occur at the initial assessment prior to beginning the intervention and after the 12-week intervention.
  Interventions: Behavioral: Integrative Cognitive Behavioural Therapy
- Wait List Control Group (No Intervention): The group do not receive the intervention and are told that they can start the intervention after 12 weeks. The participants in this group are required to complete self-reported questionnaires assessing: anxiety, depression, stress and quality of life. They are also required to attend a scalp assessment and undergo a blood test and medical photography. These assessments occur at the initial assessment prior to beginning the intervention and after the 12-week waiting period. After this 12-week waiting period, they are offered the individual therapy and their data is added to the experimental group data.

INTERVENTIONS:
Behavioral: Integrative Cognitive Behavioural Therapy — This intervention involves the psychological intervention of Cognitive Behavioural Therapy. This intervention also includes third wave psychological interventions of Mindfulness and Narrative Therapy which has been found to be helpful for people with chronic health conditions and chronic skin conditions.
  Arms: Integrative Cognitive Behavioural Therapy Intervention Group

SUMMARY:
This Randomised Control Trial (RCT) aims to test a novel Alopecia-tailored, protocolled, integrative individual psychological intervention offered to patients with enduring Alopecia. The pilot study aims to assess the impact of the intervention on 8 patients, by assessing changes in their psychological and physical symptoms (stress, anxiety, depression, quality of life, scalp hair, and other bio-markers) compared to 7 patients in the wait-list control group.

DETAILED DESCRIPTION:
Alopecia is a stress-related auto-immune skin condition that results in hair-loss on the scalp and around the body. This pilot RCT aims to test a newly developed Alopecia-specific, psychological intervention with 8 patients diagnosed with enduring Alopecia. The intervention is an Integrative Cognitive Behavioural Therapy, implemented through a protocolled programme entailing 12 weeks of hourly individual sessions. The trial will be delivered at The Dermatology Department at the Royal Free Hospital in Hampstead, London. The pilot study aims to evaluate the impact of the intervention on patients' psychological and physical symptoms (stress, anxiety, depression, quality of life, scalp hair, and other bio-markers) compared to the wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alopecia received by medical profession over 1 year prior to beginning trial
* Fluent in Written and Verbal English

Exclusion Criteria:

* Another more dominant skin condition
* Another more dominant severe and enduring mental illness
* Women who are pregnant
* Learning difficulties, brain injuries or dementia
* Drug and alcohol dependency
* Received therapy in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Other
Enrollment: 15 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety And Depression Scale (HADS) | 12 weeks
  Psychological Measure: Self-reported questionnaire assessing anxiety and depressive symptoms
Perceived Stress Scale (PSS) | 12 weeks
  Psychological Measure: Self-reported questionnaire measuring perceived stress
Dermatology Life Quality Index (DLQI) | 12 weeks
  Psychological Measure: Self-reported questionnaire measuring impact of Alopecia on participants quality of life
Severity of Alopecia Tool (SALT) Scalp Assessment | 12 weeks
  Physical Measure: Percentage of total hair loss
Blood Test | 12 weeks
  Physical Measure: Thyroid Stimulating Hormone Serum (Munit/ L) and Ferritin Serum (Micrograms)

SECONDARY OUTCOMES:
Physical Measures | 12 weeks
  Medical Photography

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hart, Doctorate, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No